CLINICAL TRIAL: NCT03923595
Title: The Puglia HCV Micro-elimination in People With Substance Use Disorders
Brief Title: Puglia HCV Micro-elimination Program
Acronym: PHCVM
Status: Completed | Type: Observational
Sponsor: Alessandra Mangia (Other)
Responsible Party: Sponsor-Investigator, Alessandra Mangia, Chief of Liver Unit, Casa Sollievo della Sofferenza IRCCS
Organization: Casa Sollievo della Sofferenza IRCCS (Other)
Other Study IDs: 19
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum of patients undergoing HCV treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adherence intervention research — dedicated management

SUMMARY:
High rates of HCV infections occur in individuals with Substance Use Disorder (SUD), particularly in subjects with Alcohol Use Disorder and in People Who Inject Drugs (PWID), but also in subjects taking psychiatric medications. In our geographic area, HCV prevalence data are available for PWID only, with >25% of them infected with HCV. The best strategy to achieve micro-elimination is targeted active screening. In Italy, SERDs assess and manage SUD individuals, but are not allowed to treat patients. Moreover, they have limited resources to perform HCV screening and to ensure linkage to care for SUD individuals living in peripheral areas. Fifteen SERDs are present in Northern Puglia and Molise, a geographical area of about 7500 Km2 usually served by our Hepatology Unit. This geographic area is not very well served by public transport leading to a logistical barrier to access needed services delivered by our unit. This issue can negatively affect engagement with clinical services for viral hepatitis even in the era of DAA. Moreover, during treatment, it is not infrequent for patients to discontinue therapy due to a chaotic lifestyle, poor income conditions and the limited access to public transportation which is needed to adhere to on-treatment monitoring. Primary objective to plan and deliver a program of dedicated transportations and cure for patients with SUD and hepatitis C who live in peripheral areas of our region. It will translate in higher rates of screening, successful linkage to care, commencement and completion of DAA treatments leading to HCV microelimination. We plan to expand our collaborative work involving up to 15 SERDs form Northen of Puglia. The program consists of -peer to peer meetings with SERDs physicians and teams, educational campaigns for patients and screening of SUD individuals and their partners using oral Quick HCV test at each SERD, - dedicated transportation services, - complete virological and liver disease evaluation at our Hospital. This organization will guarantee direct connections between Hospital and patients included in the program. This program will ensure screening of patients with suspected infection at SERD, linkage to care of newly diagnosed subjects and completion of treatment for subjects who need to start DAA therapy. The rate of screening and successful linkage to care for each SUD subgroup will be characterized as well as the cascade to care.

DETAILED DESCRIPTION:
Scientific Rationale: To adhere to the WHO plan of identifying 90% and treat 80% of HCV infected subjects, in several Countries a number of barriers need to be overcome (1). A focused effort from physicians and public administrative authorities is required to increase HCV treatment rates using direct acting antivirals (DAAs). Consequently, methods enhancing the epidemiological impact of HCV treatment using DAAs are of primary importance in order to promote what has been defined as micro-elimination (2). Among populations at high risk of transmission, targeted in the context of developing micro-elimination, people who inject drugs (PWID) and, in general, subjects with substance use disorders (SUD) are particularly important to treat.

In Italy, individuals with SUD including people who inject drugs and subjects taking psychiatric medications or alcoholic excess represent the most important target of HCV micro-elimination. Data provided by the Italian National Institute of Health during 2017, show a decline in the incidence of acute HCV infection with a peak of 0.3 x 100.000 inhabitants among subjects of 25-34 years as a consequence of: recent or ongoing use of intra venous (i.v.) substances; and/or sexual transmission (3). Moreover, in the National Cohort Piter including 9.040 HCV infected subjects, 32% was or is currently using alcohol and about 20% was or is currently using substances (4). Of interest, while alcohol abuse is usually associated with cirrhosis, drug use is associated with any stage of fibrosis. These epidemiological data highlight the need to differentiate and personalize the approach to SUD people. Finally, it is important to mention that a decline in the rate of screening has recently been registered in Italy among subjects followed by Outpatient Services for substance use disorders called SERDS (5-6). Current estimates suggest that, in our region, about 4500 subject using substances are probably HCV infected (6). Although it seems that no more than 10% of regular SERDS patients have not yet been screened for viral infections the rate of unscreened people is increasing among young SERDS patients (7). A high rate of unscreened SUD partners and families has been reported by SERDS specialists in our geographical area (personal communications).

In our real life experience only 50% of SUD patients testing HCV RNA positive agree to be treated due to different reasons including fear of treatment and difficulties in reaching DAAs treatment prescribing centers (8). Furthermore, in recent real world study leaded by our center and involving 20 out of 31 of the authorized prescribing centers in Puglia, we observed a 3% higher rate of treatment discontinuation in this, versus general population (8).

Rapid and cost-effective interventional strategies may favor both diagnosis of unknown cases and access to treatment for eligible patients. In general, training and education for providers, and an increased awareness of new advanced DAAs therapies among key risk populations are activities to strengthen within the Health system. However, in given situations, diversifying services and ensuring geographically and culturally appropriate services may play a key role in increasing the screening-diagnosis-referral-treatment-follow up cascade. It is important to establish upfront, within the heath care physicians, what can be done by different figures: the prescriber gastroenterologist is allowed to prescribe DAA and able to manage patients with a very advanced disease or patients with multiple drug-to-drug interactions; and the specialists working at the SERD are not allowed to prescribe DAA but used to monitor SUD patients and to help them to recover from their disorders.

Hypothesis: In Italy, SERDS are spread over the regional areas. According to the geographical characteristics of Puglia and Molise, the region bordering Puglia to the north, there are peripheral areas either along the cost or in internal mountains not well served by the public transportation. This aspect results in the need of relying on a private car to reach the specialized center where patients can be screened, diagnosed and treated. Fifteen SERDS are present in Northern Puglia and Molise over an area of 7500 Km2 usually served by our Hepatology Unit.

Our hypothesis is that, in addition to the known barriers to care for SUD population, lack of direct and efficient public transport represents a limitation preventing SUD individuals not only from being screened, diagnosed and treated, but also adequately informed on the most recent and highly efficient and safe pan-genotypic regimens with low impact drug to drug interactions. Moreover, the chaotic lifestyle and the poor income conditions of these patients prevent treatment completion due to transportation issue, for those who start treatment.

Primary Objective: the primary aim of this project is to explore our hypothesis by evaluating the impact of intensifying screening, diagnosis, linkage to care and treatment cascade of SUD patients through a dedicated cure program including "ad hoc" transportation.

Secondary aims are: firstly, to increase the awareness on HCV infection and related liver disease through a peer-to-peer educational campaign performed at SERDs in combination with our Unit. (Risk and liver disease outcomes, diagnostic and staging tools and the new DAAs regimens will be explained either to patients or to local healthcare workers and nurses at each individual SERD). Secondarily, to reduce treatment discontinuation in the subgroup of PWID patients.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients from SERD of 18 yrs or older either naive or previously treated including HBsAg positive and HIV positive.

Exclusion Criteria:

* GFR < 50 ml/min, pregnancy, breast-feeding, cirrhosis of CHILD-PUGH-TURCOTTE B7 o >.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV infected patients subjects with substance use disorders (SUD)
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change of linkage to care and treatment of SUD patients with HCV infection | 15 months
  to link to care a minimum of 80% of those with HCV RNA positive results as in our past experience only 50% of SUD patients positive started treatment in our area.

SECONDARY OUTCOMES:
Change of discontinuation rates of SUD patients with HCV infection | 15 months
  To reduce the rate of treatment discontinuation for SUD who start treatment, from 3% to 1.5%

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandra Mangia, San Giovanni Rotondo, Fg, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiessing L, Ferri M, Grady B, Kantzanou M, Sperle I, Cullen KJ; EMCDDA DRID group; Hatzakis A, Prins M, Vickerman P, Lazarus JV, Hope VD, Mathei C. Hepatitis C virus infection epidemiology among people who inject drugs in Europe: a systematic review of data for scaling up treatment and prevention. PLoS One. 2014 Jul 28;9(7):e103345. doi: 10.1371/journal.pone.0103345. eCollection 2014. PMID 25068274
- [Background] Mangia A, Losappio R, Cenderello G, Potenza D, Mazzola M, De Stefano G, Terreni N, Copetti M, Minerva N, Piazzola V, Bacca D, Palmieri V, Sogari F, Santoro R. Real life rates of sustained virological response (SVR) and predictors of relapse following DAA treatment in genotype 3 (GT3) patients with advanced fibrosis/cirrhosis. PLoS One. 2018 Jul 31;13(7):e0200568. doi: 10.1371/journal.pone.0200568. eCollection 2018. PMID 30063745
- [Background] Kondili LA, Vella S; PITER Collaborating Group. PITER: An ongoing nationwide study on the real-life impact of direct acting antiviral based treatment for chronic hepatitis C in Italy. Dig Liver Dis. 2015 Sep;47(9):741-3. doi: 10.1016/j.dld.2015.05.022. Epub 2015 Jun 7. No abstract available. PMID 26138800
- [Result] Lazarus JV, Safreed-Harmon K, Thursz MR, Dillon JF, El-Sayed MH, Elsharkawy AM, Hatzakis A, Jadoul M, Prestileo T, Razavi H, Rockstroh JK, Wiktor SZ, Colombo M. The Micro-Elimination Approach to Eliminating Hepatitis C: Strategic and Operational Considerations. Semin Liver Dis. 2018 Aug;38(3):181-192. doi: 10.1055/s-0038-1666841. Epub 2018 Jul 9. PMID 29986353
- [Derived] Mangia A, Rina MF, Canosa A, Piazzolla V, Squillante MM, Agostinacchio E, Cocomazzi G, Visaggi E, Augello N, Iannuzziello C, Falcone M, De Giorgi A, Campanozzi F. Increased Hepatitis C virus screening, diagnosis and linkage to care rates among people who use drugs through a patient-centered program from Italy. United European Gastroenterol J. 2021 Dec;9(10):1109-1118. doi: 10.1002/ueg2.12156. Epub 2021 Oct 26. PMID 34697911